CLINICAL TRIAL: NCT04834518
Title: Screening for Islet Autoantibodies in the Israeli Paediatric General Population for Detection of Pre-symptomatic Type-1 Diabetes Mellitus
Acronym: ADIR
Status: Recruiting | Type: Observational
Sponsor: Rabin Medical Center (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 018620RMC & 18420COM
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Type1diabetes
Keywords: autoantibodies screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Negative result at the first autoantibodies screening test: Participants will be invited to repeat the screening test at the age of 2-5 years old
- Positive result at the first or second autoantibodies screening test: * Participants will be monitored annually for risk of type 1 diabetes. (HbA1c, repeated OGTT, monitoring of urine and blood glucose where indicated)
  * Families will attend diabetes-educational program emphasizing on DKA prevention
  * Stress assessment for the families involved and stress alleviating interventions when required.

SUMMARY:
A national screening program for children aged 9 months-5 years that will be tested for the presence of islet autoantibodies.Up to 50,000 Children will be screened by their primary care physician all over Israel. The initial screening will be done at the age of 1 year (in conjunction with the routinely collection of blood for CBC ) and repeated at ages 2-5 years. Antibodies will be measured in capillary blood samples using the Ultrasensitive Antibody Detection by Agglutination-PCR (ADAP) technology developed by Enable Biosciences, which is 1,000-10,000 times more analytically sensitive than currently used methods. By using this innovative technology in such a large cohort, the study is anticipated to detect antibodies at an unprecedented earlier age.When positive in the screening, multiple antibodies will be confirmed by a second sample analyzed by the ADAP technology. In addition, multiple antibodies will be also measured using a radio-binding assay (RBA) of a venous blood sample for investigational purpose only. Children with confirmed multiple antibodies (stage 1 or 2 T1D) will be followed up routinely for the appearance of clinical signs of diabetes (HbA1c, repeated OGTT, monitoring of urine and blood glucose where indicated) and will be invited along with their families to attend an educational program. This program will include diabetes education emphasizing on DKA prevention as well as stress assessment for the families involved and stress alleviating interventions. The analysis and storage of the samples will be done in a single screening center at Schneider Children's Medical Center of Israel.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Children aged 9-months- 5 years at first screening.

Exclusion Criteria:

* Known diagnosis of diabetes (Type 1 or other)

Ages: 9 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from the general population of all over Israel, aged 9 months-5 years arriving to the routine blood test for CBC or to any other routine visit to the community pediatrician.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of presymptomatic type 1 diabetes | End of screening and follow-up period-4 years after obtaining the first screening test
  Presymptomatic type 1 diabetes, defined as positive for 2 or more islet autoantibodies (GADA, IA-2A, and IAA) or those with high levels of a single antibody in both the screening and confirmation samples or in the screening sample plus a diagnosis of diabetes prior to obtaining the conformation sample.
  Presymptomatic type 1 diabetes will be classified as stage 1, 2, or 3:
  * Stage 1 will be defined as 2 or more islet autoantibodies or high levels of a single antibody and normal glucose tolerance based on OGTT results. (not including patients with only a single antibody who have first degree relative with type 1 diabetes)
  * Stage 2 will be defined as 1 or more islet autoantibodies accompanied by dysglycemia (fasting plasma glucose of 110-125 mg/dL or impaired 2-hour plasma glucose of 140- 199 mg/dL and/or plasma glucose ≥200 mg/dL at intermediate time points [30, 60, 90 minutes]) based on OGTT results.
  * Stage 3 will be defined according to the American Diabetes Association criteria
Frequency of Diabetic Ketoacidosis on the clinical presentation of Type 1 Diabetes | End of screening and follow-up period-4 years after obtaining the first screening test

SECONDARY OUTCOMES:
The average age of islet autoantibody seroconversion | End of screening and follow-up period-4 years after obtaining the first screening test
The rate of islet autoantibody seroconversion | End of screening and follow-up period-4 years after obtaining the first screening test
The rate of progression from pre-symptomatic T1D to clinical diabetes | End of screening and follow-up period-4 years after obtaining the first screening test

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Study Director — Schneider Children's Medical Center
Locations (7):
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah medical Center, Jerusalem
  - Child Health Centers all over Israel (clalit Health Services), Petah Tikva
  - Schneider Children Medical Center of Israel, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Dana-Duek children's hospital, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided